CLINICAL TRIAL: NCT06029309
Title: A Phase 1/2 Study of Zanubrutinib and Tafasitamab in Mantle Cell Lymphoma
Brief Title: Zanubrutinib and Tafasitamab in Mantle Cell Lymphoma
Acronym: ZANU-TAFA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alvaro Alencar, MD (Other)
Collaborators: BeiGene (Industry); Incyte Corporation (Industry); MorphoSys AG (Industry)
Responsible Party: Sponsor-Investigator, Alvaro Alencar, MD, Associate Professor of Clinical, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20221346
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — zanubrutinib; tafasitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zanu-Tafa Phase 1 Group (Experimental): Participants in this group will receive combination therapy of Zanubrutinib (Zanu) and Tafasitamab (Tafa) for up to 24 cycles, followed by maintenance therapy with Zanubrutinib until progression. Each cycle is 28 days in length. Combination therapy will be administered via induction phases as follows:
  1. Early induction - cycles 1 to 3 (12 weeks)
  2. Late induction - cycles 4 to 12 (36 weeks)
  3. Extended induction - cycles 13-24 (48 weeks)
  Subsequent maintenance Zanu therapy may last up to 2 years. Total study participation is up to four (4) years.
  Interventions: Drug: Zanubrutinib; Drug: Tafasitamab
- Zanu-Tafa Phase 2 Group (Experimental): Participants in this group will receive the combination therapy of Zanubrutinib (Zanu) at the recommended phase 2 dose (RP2D) determined during Phase 1, and Tafasitamab at standard doses, followed by maintenance therapy with Zanubrutinib until progression.. Combination therapy will be administered via induction phases as follows:
  1. Early induction - cycles 1 to 3 (12 weeks)
  2. Late induction - cycles 4 to 12 (36 weeks)
  3. Extended induction - cycles 13-24 (48 weeks)
  Subsequent maintenance Zanu therapy may last up to 2 years. Total study participation is up to four (4) years.
  Interventions: Drug: Zanubrutinib; Drug: Tafasitamab

INTERVENTIONS:
Drug: Zanubrutinib — Participants will be administered Zanubrutinib orally (PO) via capsules daily during each 28-day cycle at the following dose levels:
  * Phase 1 Dose Level 1: 320 mg
  * Phase 1 Dose Level -1: 240 mg
  * Phase 2: Recommended dose determined in Phase 1.
Drug: Tafasitamab — Participants will be administered a 12 mg/kg dose of Tafasitamab intravenously (IV) during each 28-day cycle as follows:
  * Early Induction - Cycle 1: Days 1, 4, 8, 15, and 22
  * Early Induction - Cycles 2 and 3: Days 1, 8, 15 and 22
  * Late Induction - Cycles 4 through 12: Days 1 and 15

SUMMARY:
The main purpose of this study to find the ideal dose for the combination treatment of Zanubrutinib and Tafasitamab in patients with mantle cell lymphoma. Another purpose is to assess how well the combination treatment works in patients with the study disease.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age
2. Patients must have histologic confirmation of mantle cell lymphoma (MCL) defined by the World Health Organization (WHO) classification
3. Baseline PET/CT scans must demonstrate fluorodeoxyglucose (FDG) avid lesions compatible with CT defined anatomical tumor sites. Patients should have at least one measurable site of disease per Lugano classification
4. Patient should have indication according to primary investigator for treatment initiation
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
6. Life expectancy of greater than 4 months.
7. Willingness to avoid pregnancy or fathering children during the study and for at least 90 days after the last dose of the study drug.
8. Patients must have normal organ and marrow function as defined below:

   1. Absolute neutrophil count >1,000/mm3 independent of growth factor support within 7 days of study entry (>700/mm3 if lymphoma involvement of the bone marrow or spleen)
   2. Platelets >70,000/mm3 independent of transfusion support within 7 days of study entry (>50,000/mm3 independent of transfusion support within 7 days of study entry if lymphoma involvement of the bone marrow or spleen)
   3. Hemoglobin >9 g/dL or >8 g/dL in case of bone marrow involvement by lymphoma independent of transfusion support within 7 days of study entry.
   4. Total bilirubin < 1.5 x within normal institutional limits (unless known history of Gilbert's disease or up to 3 x upper limit of normal (ULN) if due to lymphoma involvement of liver)
   5. Gamma-Glutamyl Transpeptidase (GGT)/Aspartate transaminase (AST, SGOT)/Alanine transaminase (ALT, SGPT) ≤ 2.5 x institutional upper limit of normal
   6. Creatinine within normal institutional limits, or creatinine clearance ≥ 40 mL/min (as estimated by the Cockcroft-Gault equation) for patients with creatinine levels above institutional normal (creatinine clearance ≥ 30 mL/min as estimated by the Cockcroft-Gault equation if due to lymphoma).

Inclusion Criteria, Phase 1 Only:

1. Relapsed MCL patients with at least 1 but no more than 3 lines of therapy, regardless of previous Bruton Tyrosine Kinase (BTK) inhibitor exposure

Inclusion Criteria, Phase 2 Only:

1. Untreated symptomatic MCL deemed by the primary investigator not to be eligible for intensive combination immunochemotherapy.

Exclusion Criteria, Phase 1 and 2:

1. Patients receiving any other investigational agents
2. Patients with known central nervous system involvement of lymphoma
3. Uncontrolled intercurrent illness such as: clinically significant active cardiovascular disease such as uncontrolled or symptomatic arrhythmia, uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) Class III-IV, history of myocardial infarction within 6 months of screening, stroke in last 6 months, liver cirrhosis, autoimmune disorder requiring immunosuppression or long-term corticosteroids (>10 mg daily prednisone equivalent), or any other serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
4. QT interval corrected with Fridericia's formula (QTcF) > 450 msec or other significant ECG abnormalities including second-degree atrioventricular block Type II, or third-degree atrioventricular block
5. Prior or concurrent malignancies with exception of surgically cured carcinoma in situ (CIS) of the uterus, carcinoma of the skin without evidence of disease for ≥5 years
6. Concurrent malignancy requiring active therapy
7. Known seropositive and requiring anti-viral therapy for human immunodeficiency virus
8. Breastfeeding or pregnant women
9. Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody will need a polymerase chain reaction (PCR) below cutoff value prior to enrollment. (PCR positive patients will be excluded). Hepatitis C antibody positive patients are eligible if PCR is negative. Hepatitis B core antibody (+) patients without evidence of HBsAg or Hep B PCR (+) are eligible with appropriate Hepatitis B reactivation prophylaxis
10. Ongoing treatment with medications that are moderate or strong cytochrome P (CYP) 450, family 3, subfamily A (CYP3A) inhibitors, or strong CYP3A inducers that cannot be safely substituted. For patients with ongoing treatment with these medications that can be safely substituted, minimum washout period should be 7 days or five half-lives, whichever is shorter.
11. History of allogenic hematopoietic stem cell transplantation prior to enrollment
12. Active systemic infection (including severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) positive test) or other Active infection including infections requiring oral or intravenous antimicrobial therapy.
13. Administration of live vaccine within 28 days prior to start of study treatment
14. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the patient's safety or put the study at risk.
15. Toxicity must have recovered to ≤ Grade 1 from prior chemotherapy (except for alopecia, absolute neutrophil count, and platelet count). (Please refer to Inclusion Criteria 7 and 8 for absolute neutrophil count and platelet count, respectively.)
16. Unable to swallow capsules, or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
17. Prior corticosteroids in excess of prednisone 10 mg/day or its equivalent with antineoplastic intent within 7 days of the start of study drug. Prior chemotherapy, targeted therapy, or radiation therapy within 3 weeks, antineoplastic therapy with Chinese herbal medication or antibody-based therapies within 4 weeks of the start of study drug.
18. History of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention
19. History of stroke or intracranial hemorrhage within 180 days before first dose of study drug
20. Major surgery within 4 weeks of the first dose of study drug
21. Patient requires treatment with warfarin or other vitamin K antagonists
22. Any contraindication per Tafasitamab United States Prescribing Information (USPI).
23. Patients with impaired decision-making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2032-05-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Recommended Phase 2 Dose (RP2D) of Zanubrutinib | 4 weeks
  Determination of the RP2D of Zanubrutinib, when used in combination with Tafasitamab, based on evaluation of dose limiting toxicity (DLT) in participants during the Phase 1 part of the study. DLT will be defined as the occurrence of specified adverse events (AEs) at least possibly related to the study therapy during the DLT review period.
Phase 2: Rate of Complete Response (CR) to Zanubrutinib at RP2D | Up to 48 weeks
  The complete response (CR) rate among study participants in Phase 2 to Zanubrutinib at the RP2D in combination with Tafasitamab will be assessed. Response will be assessed using positron emission tomography (PET)/computerized tomography (CT) according to the Lugano 2014 criteria. CR will be defined by a Deauville score of less than or equal to (≤) 3.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 48 weeks
  The overall response rate (ORR) in study participants will be assessed. ORR will be defined at the percentage of participants achieving complete response (CR) or partial response to study therapy at at the end of early (cycles 1-3) and late induction (cycles 4-12). Response to treatment will be assessed using PET/CT according to Lugano 2014 criteria after weeks 12 and 48 of treatment. CR will be defined by a Deauville score of ≤ 3, and PR by a Deauville score of 4 or 5 with reduced uptake from baseline.
Progression-free Survival (PFS) | Up to 48 months
  Progression-free survival among study participants will be assessed during treatment and clinical follow-up. PFS is defined as the time from start of treatment until disease progression or death.
Overall Survival (OS) | Up to 48 months
  Overall survival (OS) among study participants will be assessed during treatment and clinical follow-up. OS is defined from start of treatment until death from any cause.
Number of Participants Experiencing Treatment-related Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 27 months
  The dosing, safety, and feasibility of combination of Zanubrutinib and Tafasitamab will be assessed and reported among study participants in Phase 1 as the number of participants experiencing treatment-related toxicity after start of study therapy, including treatment-related adverse events (AEs) and serious adverse events (SAEs). AEs and SAEs will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5, per physician discretion.
Phase 2: Duration of Response (DOR) | Up to 48 months
  The duration of response (DOR) among study participants will be assessed during treatment and clinical follow-up. DOR is defined as the time from randomization to disease progression or death in patients who achieve complete response (CR) or partial response (PR).
Phase 2: Time to Next Treatment (TTNT) | Up to 24 months
  Time to next treatment (TTNT) is defined as the time between the date of initiation of proposed treatment and the date of next subsequent systemic treatment initiation. For participants who do not have a subsequent treatment, the TTNT will be censored at last date known to be alive, except that death from any cause will be considered a competing risk event.

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Alencar, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No